CLINICAL TRIAL: NCT04188626
Title: Identification of Physiological and Behavioural Biomarkers to Predict Take-over Control Quality in Level 3 Conditionally Automated Vehicles
Brief Title: Identification of Biomarkers to Predict Driver Take-over Control Quality
Acronym: ANTIDOTE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PSA Automobiles S.A. (Industry)
Collaborators: University of Bordeaux (Other); University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: XP THSE BDX SNPSY; ID-RCB (ANSM number) (Other: 2019-A01524-53)
Record Dates: First submitted 2019-11-18; First posted 2019-12-06 (Actual); Last update posted 2020-09-21 (Actual); Status verified 2020-09

CONDITIONS: Healthy Subjects; Attention Deficit
Keywords: Automated driving; Conditional automation; Driver distraction; Driver take-over quality; Biomarkers
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Intervention Model Description: Monocentric preliminary study including an experimental driving session in a driving simulator.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Driving session (Experimental): The volunteers will be placed in a driving simulator that will simulate autonomous highway driving.
  Interventions: Behavioral: Driving simulator sessions

INTERVENTIONS:
Behavioral: Driving simulator sessions — The volunteers will be placed in a driving simulator that will simulate autonomous highway driving. This autonomous driving will be interrupted by take-over requests related to events that disrupt autonomous driving. During autonomous driving, the driver will have to disengage from driving by performing non-related driving tasks. During each non-related driving tasks, a take-over request will be sent. Electrophysiological (EEG, ECG, EDA, EMG, respiration) and behavioural data will be recorded before, during and after the take-over control.

SUMMARY:
At level 3 conditionally automated, the vehicle ensures driving and the driver disengages from driving to perform another activity independent of driving (ex: read a book, play on his phone ....). However, drivers are expected to be available to take over control for the case of system failure or limitation. This take-over control must take place in a limited time, very short, of the order of a few seconds. To take-over control of the vehicle quickly and efficiently, the driver must be, at the time of take-over, vigilant, efficient, and attentive to the environment and focused on the take-over of manual driving. Predicting the driver's reengagement capabilities to ensure that the driver will be able to take-over control of the vehicle is crucial at level 3 of autonomous driving.

The objective of ANTIDOTE is to determine physiological and behavioural parameters capable of predicting the take-over quality in level 3 conditionally automated vehicles in a simulated highway driving situation in healthy drivers or drivers with attention disorders.

DETAILED DESCRIPTION:
At level 3 conditionally automated, the vehicle ensures driving and the driver disengages from driving to perform non-related driving tasks (ex: read a book, play on his phone ....). However, drivers are expected to be available to take over control for the case of system failure or limitation. This take-over control must take place in a limited time, very short, of the order of a few seconds. To take-over control of the vehicle quickly and efficiently, the driver must be, at the time of take-over, vigilant, efficient, and attentive to the environment and focused on the take-over of manual driving. Predicting the driver's reengagement capabilities to ensure that the driver will be able to take-over control of the vehicle is crucial at level 3 of autonomous driving.

In this context, the objective of ANTIDOTE is to determine physiological and behavioural parameters capable of predicting the take-over quality in level 3 conditionally automated vehicles in a simulated highway driving situation.

This study will examine how engagement will impact take-over control quality in 6 non-driving related secondary tasks. A driving simulator study will be conducted and data from a total of 32 healthy drivers and 16 drivers with attention disorders will be used to evaluate take-over quality.

Electrophysiological (EEG, ECG, EDA, EMG, respiration) and behavioral data will be recorded before, during and after the take-over control.

ELIGIBILITY:
Inclusion Criteria:

Common inclusion criteria:

* male or female aged between 20 and 75 years old
* BMI between 18 and 27
* Subject size between 1.50 m and 1.95 m
* Without sleep complains (Item of Basic Nordic Sleep Questionnaire ≤ 3)
* Without excessive daytime sleepiness (Epworth score ≤ 11)
* Non-professional drivers
* Subjects with a driver's license for at least one year
* Subjects driving at least 5000 km per year.
* Having normal visual acuity (correction with lenses accepted) and normal color vision
* Affiliated to a national health service
* Having given written informed consent to participate in the trial.

Healthy volunteers specific inclusion criteria:

* SCL90R score < 60 for anxiety and depression subscales
* MMSE ≥ 30

ADHD patients specific inclusion criteria:

* Patients with an ADHD disorder according to DSM 5,
* Patients agreeing to discontinue psychostimulant treatment 48 hours prior to the experimental session,

Exclusion Criteria:

* Severe life-threatening conditions in the short term,
* Unstable endocrine diseases
* Progressive cardiovascular diseases
* Progressive neurological diseases treated or not,
* Addiction to a substance
* Night and shift-workers who has taken a constraints in the last 72 hours,
* Psychotropic medication taking
* Benzodiazepine or Z-drug medication taking
* Cardiotropic medication taking
* Volunteers who need glasses to drive
* Having simulator-sickness during the first practice session

Healthy volunteers specific inclusion criteria:

* Psychiatric co-morbidities: current major depressive episode, current hypomanic or manic episode, psychotic disorders, autism spectrum disorder
* Exceeded consumption of coffee, tea or caffeinated drinks(> 5 cups / day)
* Exceeded consumption of alcohol drinks (> 2 drinks / day during the last 6 months)

ADHD patients specific inclusion criteria:

* Psychiatric co-morbidities: current major depressive episode, current hypomanic or manic episode, psychotic disorders, autism spectrum disorder (except ADHD)
* Exceeded consumption of alcohol drinks(> 3 drinks / day during the last 6 months)

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2019-12-09 (Actual); Primary Completion 2020-08-06 (Actual); Study Completion 2020-08-06 (Actual)

PRIMARY OUTCOMES:
Quality of driving take-over behaviour | 8 secondes after take-over request
  Quality of driving take-over behaviour (Good/bad) will be assessed by collision (collision or driving off the road) and critical encounters (Time To Collision).
  Time to collision (TTC) refers to the time required for the vehicle to collide with the stationary obstacle obstructing the driving lane if it continues at its speed at the time it changes to the next lane completely.
  Good : no collision AND TTC >= 1.5 secondes Bad : collision or no collision AND TTC < 1.5 secondes

SECONDARY OUTCOMES:
EEG (electroencephalogram) | during the 2 minutes before the take-over request, during take-over control and the 2 minutes after the take-over control
  Physiological parameter: EEG will be recorded and Alpha, theta and gamma activity will be analyzed in the waking EEG.
ECG (electrocardiogram) | during the 2 minutes before the take-over request, during take-over control and the 2 minutes after the take-over control
  Physiological parameter : ECG recordings and heart rate variability based on time and frequency domain will be analyzed.
EMG (electromyogram) | during the 2 minutes before the take-over request, during take-over control and the 2 minutes after the take-over control
  Physiological parameter : surface EMG will be recorded and Derive Average Rectified, derive Integrated Root and means Square EMG will be analyzed and EMG Frequency & Power Analysis.
Electrodermal activity 1 (EDA) | during the 2 minutes before the take-over request, during take-over control and the 2 minutes after the take-over control
  Physiological parameter : EDA will be recorded and skin conductance level analyzed.
Electrodermal activity 2 (EDA) | during the 2 minutes before the take-over request, during take-over control and the 2 minutes after the take-over control
  Physiological parameter : EDA will be recorded and skin conductance response analyzed.
Respiration | during the 2 minutes before the take-over request, during take-over control and the 2 minutes after the take-over control
  Physiological parameter : Respiratory frequency recorded
Physical activity | during the 2 minutes before the take-over request, during take-over control and the 2 minutes after the take-over control
  Physiological parameter : Physical activity expressed in count/min
Eye tracking | during the 2 minutes before the take-over request, during take-over control and the 2 minutes after the take-over control
  Physiological parameter :Eye tracking will be recorded and point of gaze, Perclos, blinks, diameters of pupils analyzed.
Subjective driving take-over control quality: Visual analogic scale | 8 secondes after take-over request
  Visual analogue scale to assess subjective driving take-over control quality (Subjective scale).
  The scale ranges from 0 " bad" to 100 "good"
Subjective level of attention and distraction before take-over control request | 8 secondes after take-over request
  Visual analogue scale to assess subjective level of attention and distraction just before take-over control request The scale ranges from 0 "attentive" to 100 "inattentive"

CONTACTS AND LOCATIONS:
Overall Officials: Pierre PHILIP, MDPhD, Principal Investigator — Bordeaux University Hospital - Bordeaux University
Locations (1):
- Bordeaux University Hospital, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No
Patient could request investigator or Data Protection Officer an access to IPD according to French regulation (act No. 78-17 of 6 January 1978 on data processing, data files and individual liberties, amended by act No. 2004-801 of 6 August 2004) and he EU General Data Protection Regulation (GDPR) of 27 april 2016 applicable since 25 May 2018.